CLINICAL TRIAL: NCT05988125
Title: Prospective Registry Study of Endovascular Treatment for Acute Ischemic Stroke Patients in China
Brief Title: Prospective Registry Study of Endovascular Treatment for Acute Ischemic Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tingyu-Yi (Other)
Collaborators: Fujian Medical University Union Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); First People's Hospital of Shenyang (Other)
Responsible Party: Sponsor-Investigator, Tingyu-Yi, Prospective Registry Study of Endovascular Treatment for Acute Ischemic Stroke Patients in China, Zhangzhou Municipal Hospital
Organization: Zhangzhou Municipal Hospital (Other)
Other Study IDs: ETERNITY
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-01

CONDITIONS: Endovascular Treatment
Keywords: acute Ischemic Stroke; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To investigate the real situation of assessment, diagnosis and treatment of acute ischemic stroke patients with endovascular therapy.

DETAILED DESCRIPTION:
Prospective Registry Study of Endovascular Treatment for Acute Ischemic Stroke Patients is an academic,independent, pragmatic , prospective, multicenter, observational registry study. The acute ischemic stroke patients undergone endovascular therapy will be enrolled in stroke centers. Baseline information and clinical follow-up information at 90 days of stroke onset are collected. Data collected include demographics, comorbidities, pathogenesis, blood pressures, stroke severity on admission, time intervals, reperfusion condition, and functional outcome, et al. The study aims to investigate the real situation of assessment, diagnosis and treatment of acute ischemic stroke patients with endovascular therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke;
2. Brain imaging confirmed intracranial large vessel occlusion: intracranial internal carotid artery (ICA), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA V4), and posterior cerebral artery (PCA P1);
3. Initiation of any type of endovascular treatment, including mechanical thrombectomy, aspiration, angioplasty, and stenting;
4. Informed Consent as documented by signature or fulfilling the criteria for emergency consent/ deferral consent

Exclusion Criteria:

1. Acute intracranial haemorrhage
2. No evidence of large vessel occlusion on digital subtraction angiography.
3. Patient bedridden or presenting from a nursing home
4. Foreseeable difficulties in follow-up due to geographic reasons (e.g. patients living abroad) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients receiving endovascular treatment.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score at 90 days | 90 days
  The range of the modified Rankin Scale is from 0 to 6. A higher score indicates a worse outcome.
  0-No symptoms; 1-No significant disability; 2-Slight disability; 3-Moderate disability; 4-Moderately severe disability; 5-Severe disability; 6-Dead.

SECONDARY OUTCOMES:
Successful reperfusion rate | 90 days
symptomatic intracranial hemorrhage or death within 90 days after stroke onset. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Wen-huo Chen, bachelor, Principal Investigator — Zhangzhou Affiliated Hospital to Fujian Medical University , Fujian ,China
Locations (6):
- China (6):
  - Zhangzhou Municipal Hospital, Zhangzhou, Fujian
  - Gansu provincial hospital of TCM, Lanzhou, Gansu
  - Jiamusi Central Hospital, Jiamusi, Heilongjiang
  - Department of Neurology, The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Songyuan Jilin Oilfield Hospital, Songyuan, Jilin
  - Shenyang First People's Hospital, Shenyang, Liaoning